CLINICAL TRIAL: NCT04111367
Title: A Phase IIa, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Seraprevir in Combination With Sofosbuvir in Patients With Chronic Genotype 2,3,6 Hepatitis C Virus Infection
Brief Title: Study of Seraprevir in Combination With Sofosbuvir in Chronic Genotype 2,3,6 Hepatitis C Virus Infection Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ginkgopharma CO., LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GP205-1901
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotype 2 and 6 Subjects (Experimental): Genotype 2 and 6 Subjects will receive oral tablets of Seraprevir 200mg twice a day along with oral tablet of sofosbuvir 400 mg,once a day from Day 1 up to Week 12
  Interventions: Drug: Seraprevir; Drug: Sofosbuvir
- Genotype 3 Subjects (Experimental): Genotype 3 Subjects will receive oral tablets of Seraprevir 200mg twice a day along with oral tablet of sofosbuvir 400 mg,once a day from Day 1 up to Week 24
  Interventions: Drug: Seraprevir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Seraprevir — Subjects will receive oral tablets of Seraprevir 100 mg, twice a day from Day 1 up to Week 12，the other group will receive the same dose for 24 weeks.
  Other Names: GP205
Drug: Sofosbuvir — Subjects will receive oral tablet of sofosbuvir 400 mg, once a day from Day 1 up to Week 12,the other group will receive the same dose for 24 weeks.
  Other Names: sovaldi

SUMMARY:
This study was to assess the safety and efficacy of Seraprevir in combination with sofosbuvir in patients with Hepatitis C (HCV) genotype2,3,6. Efficacy was assessed by the rate of sustained viral response (SVR) 12 weeks after the discontinuation of therapy (SVR12).

ELIGIBILITY:
Inclusion Criteria:

Hepatitis C virus (HCV) genotype 2,3,6 infection (confirmed at screening). HCV RNA greater than 10,000 IU/mL at screening. Participant must be willing and able to comply with the protocol requirements. weight was more than 40 kg. age is between 18-75,either sex.

Exclusion Criteria:

Co-infection with hepatitis B virus or human immunodeficiency virus (HIV). Infection with HCV non-genotype 2,3,6,or Infection with mixed genotype,or Genotype cannot be confirmed.

Medical history of major functional organ transplantation. Suffering from serious blood system disease(such us Thalassemia/Sickle Cell Anemia).

Participation in a clinical study within 3 months prior to first dose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Sustained Virologic Response 12 Weeks After the Actual End of Treatment（SVR12） | Posttreatment Week 12
  SVR12 is defined as HCV RNA < the lower limit of quantification (LLOQ; ie, < 15 IU/mL) 12 weeks following the last dose of study drug.

SECONDARY OUTCOMES:
Percentage of Participants Achieving a Sustained Virologic Response 4 Weeks After the Actual End of Treatment (SVR4) | Posttreatment Week 4
  SVR4 is defined as HCV RNA < LLOQ at 4 weeks following the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Xuegang Wu, Study Director — Ginkgo Pharma Co., Ltd.
Locations (4):
- China (4):
  - Beijing Ditan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Liuzhou General Hospital, Liuchow, Guangxi
  - The first hospital of JILIN University., Changchun, Jilin
  - The First Affiliated Hospital Of Guangxi Medical University, Guangxi, Nanning